CLINICAL TRIAL: NCT05479539
Title: Effects of Action Observation Therapy in Patients Undergoing Surgery for Shoulder-instability
Brief Title: Action Observation Therapy in Patients Undetgoing Surgery for Shoulder Instability
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLF21/03
Record Dates: First submitted 2022-07-27; First posted 2022-07-29 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Shoulder Instability

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AOT (Experimental)
  Interventions: Behavioral: Action observation therapy
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Action observation therapy — Participants will watch 12-minute video-clips followed by 8 minutes of motor imagery. Video-clips observation and imagination will be focused un shoulder tasks occuring on the three planes of motion.
  Arms: AOT

SUMMARY:
The study will aim at investigating the effects of action observation therapy (action observation plus motor imagery) in patients with shoulder instability undergoing capsulo-plastic surgery. Forty subjects scheduled for capsulo-plastic surgery will be randomized into an AOT or Control group. AOT group will undergo action observation followed by motor imagery of upper limb motor tasks for 4 weeks after surgery, whereas Control group will perform no intervention. In addition, both groups will undergo postoperative usual care including immobilization with a brace and passive upper limb mobilization. All participants will be assessed for shoulder pain, function, range of motion, fear of movement and quality of life the day before surgery, at training end and 3 months after training end.

ELIGIBILITY:
Inclusion Criteria:

* Subjects undergoing capsule-plastic surgery or Latarjet stabilization for shoulder instability

Exclusion Criteria:

* Previous upper limb surgery
* Cognitive impairments
* Visual or auditory impairments
* Postoperative complications limiting upper limb motor recovery (e.g., infections)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Changes in shoulder function | At baseline, after 4 weeks of training and at 3 month after the training end
  Simple shoulder test
Changes in shoulder function | At baseline, after 4 weeks of training and at 3 month after the training end
  Disability Arm Shoulder Hand - DASH

SECONDARY OUTCOMES:
Changes in shoulder pain | At baseline, after 4 weeks of training and at 3 month after the training end
  Numerical Pain Rating Scale (0 - best outcome, 100 worst outcome)
Changes in shoulder range of motion | At baseline, after 4 weeks of training and at 3 month after the training end
  Flexion, abduction, inernal and external rotation range of motion assessed using a goniometer
Changes in fear of movement | At baseline, after 4 weeks of training and at 3 month after the training end
  Tampa scale of kinesiophobia
Changes in quality of life | At baseline, after 4 weeks of training and at 3 month after the training end
  Short Form - 36 items

IPD SHARING:
Plan to Share IPD: No